CLINICAL TRIAL: NCT03050073
Title: Choroidal Thickness Association With Primary Angle Closure
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: IRIS
Record Dates: First submitted 2017-02-07; First posted 2017-02-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Choroidal Thickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A chinese study shows that chinese population eyes with a primary angle closure have a greater choroidal thickness than normal eyes.The increase of choroidal thickness would be associated to this primary angle closure.

DETAILED DESCRIPTION:
Usual ophtalmic consultation for glaucoma with primary angle closure

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Primary angle closure confirmed by gonioscopy
* interpretable images for choroidal thickness measure
* interpretable images by Ultra Bio Microscopy (UBM)

Exclusion Criteria:

* Acute crisis for angle closure
* Rethinopathy (diabetic or hypertensive)
* Histories of intra-eye surgery
* Great myopia
* Hypermetropia
* retinal pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient consulting for glaucoma or not with primary angle closure
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
change of choroidal thickness measurement by Imaging of the fundus oculi (OCT swept source) | Day 1 Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BEAUSSIER, Pharm-D, Study Director — CRC
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided